CLINICAL TRIAL: NCT02928757
Title: Complex Care for Kids Ontario (CCKO): A Patient- and Family-centred Implementation and Evaluation of Care Coordination for Children With Medical Complexity
Brief Title: Complex Care for Kids Ontario (CCKO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); London Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Eyal Cohen, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000053509
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Children With Medical Complexity
Keywords: Care coordination; Complex care kids Ontario; Technology-dependent; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): In addition to standard medical care, participants will be enrolled to be seen as soon as possible in a complex care clinic as part of the CCKO initiative.
  Interventions: Other: Complex care clinic as part of the CCKO initiative
- Wait-list Group (No Intervention): The control group will receive usual care, but will be wait-listed for 1 year to be seen in a complex care clinic as part of the CCKO initiative.

INTERVENTIONS:
Other: Complex care clinic as part of the CCKO initiative — The CCKO intervention involves intensive care coordination, defined as: "deliberate organization of patient care activities between two or more participants (including the patient) involved in a patient's care to facilitate the appropriate delivery of health care services. Organizing care involves marshaling of personnel and other resources needed to carry out all required patient care activities and is often managed by the exchange of information among participants responsible for different aspects of care". Within CCKO, intensive care coordination will specifically include: 1) the tailored, family/health care provider co-creation and regular updating of care coordination plans for each child which will be 2) facilitated and accounted for by key workers partnering with families.
  Arms: Intervention Group

SUMMARY:
There are ~6,200 children in Ontario with special and complex healthcare needs requiring multiple services from many different doctors and other healthcare providers. These children are at a high risk of missed, duplicated or inappropriate care, and extraordinary financial burden and stress on families. While small in number (<1% of Ontario kids), these children use 1/3 of all child healthcare resources, and are known to desperately need coordinated care to optimize their health. Complex Care Kids Ontario (CCKO) brings together researchers, children and families, and healthcare providers from across Ontario to develop, implement and evaluate an evidence-based and coordinated model of care for every child with medical complexity in Ontario.

ELIGIBILITY:
Inclusion Criteria (Meets at least ONE criterion from EACH of the following four conditions):

* Technology dependent and/or users of high intensity care
* Child is dependent on mechanical ventilators, and/or requires prolonged IV administration of nutritional substances or drugs and/or is to have prolonged dependence on other device-based support. For example: tracheostomy tube care/ artificial airway, suctioning, oxygen support, or tube feeding
* Child has prolonged dependence on medical devices to compensate for vital bodily functions, and requires daily/ near daily nursing care, e.g., cardiorespiratory monitors; renal dialysis due to kidney failure
* Fragility
* The child has severe and/or life-threatening condition
* Lack of availability and/or failure of equipment/technology or treatment places the child at immediate risk resulting in a negative health outcome
* Short-term changes in the child's health status (e.g., an intercurrent illness) put them at immediate serious health risk
* Chronicity
* The child's condition is expected to last at least six more months
* The child's life expectancy is less than six months
* Complexity
* Involvement of at least five healthcare practitioners/ teams and healthcare services are delivered in at least three of the following locations: Home, School/Nursing school, Hospital, Children's Treatment Centre, Community-based clinic (e.g. doctor's office), Other (at clinician's discretion)

Exclusion Criteria:

* High Utilization of hospital level care
* ≥ 3 hospitalizations, ≥ 2 ICU admissions, ≥ 30 days of total hospitalization in previous 3 months, excluding newborn admission
* Patient with tracheostomy and home ventilation
* Medical Status is deemed highly fragile and the need for close follow-up is deemed essential by both referring and triaging team
* Already followed by a complex care team
* >16.0 years of age
* Inadequate English language skills to comprehend study questionnaires

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2016-12; Primary Completion 2021-01 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Service delivery outcomes: coordination of care among health providers and families, coordination of care between health providers and families, utility of follow-up planning tools | Baseline
  These outcomes will be assessed with the Family Experiences with Coordination of Care (FECC) survey.
Service delivery outcomes: coordination of care among health providers and families, coordination of care between health providers and families, utility of follow-up planning tools | 6 months
  These outcomes will be assessed with the Family Experiences with Coordination of Care (FECC) survey.
Service delivery outcomes: coordination of care among health providers and families, coordination of care between health providers and families, utility of follow-up planning tools | 12 months
  These outcomes will be assessed with the Family Experiences with Coordination of Care (FECC) survey.
Service delivery outcomes: coordination of care among health providers and families, coordination of care between health providers and families, utility of follow-up planning tools | 24 months
  These outcomes will be assessed with the Family Experiences with Coordination of Care (FECC) survey.

SECONDARY OUTCOMES:
Child quality of life & overall emotional health | Baseline
  These outcomes will be assessed using the using the "Feelings" subscale from the KIDSCREEN-52 (6 items), used in over 250 studies in the child health services literature since its publication in 2005.
Child quality of life & overall emotional health | 6 months
  These outcomes will be assessed using the using the "Feelings" subscale from the KIDSCREEN-52 (6 items), used in over 250 studies in the child health services literature since its publication in 2005.
Child quality of life & overall emotional health | 12 months
  These outcomes will be assessed using the using the "Feelings" subscale from the KIDSCREEN-52 (6 items), used in over 250 studies in the child health services literature since its publication in 2005.
Child quality of life & overall emotional health | 24 months
  These outcomes will be assessed using the using the "Feelings" subscale from the KIDSCREEN-52 (6 items), used in over 250 studies in the child health services literature since its publication in 2005.
Child physical pain | Baseline
  Children's physical pain will be measured using only self or proxy reports of pain according to a 10 cm linear Visual Analog Scale (VAS).
Child physical pain | 6 months
  Children's physical pain will be measured using only self or proxy reports of pain according to a 10 cm linear Visual Analog Scale (VAS).
Child physical pain | 12 months
  Children's physical pain will be measured using only self or proxy reports of pain according to a 10 cm linear Visual Analog Scale (VAS).
Child physical pain | 24 months
  Children's physical pain will be measured using only self or proxy reports of pain according to a 10 cm linear Visual Analog Scale (VAS).
Parents' Quality of Life | Baseline
  Parents' quality of life will be measured according to a subjective life appraisal definition with Diener's highly validated Satisfaction with Life Scale (SWLS) (5 items) which is the most validated life satisfaction scale in health and social sciences literature.
Parents' Quality of Life | Baseline
  Parents' quality of life will also be measured with an adapted version of the KIDSCREEN survey subscale for Feelings.
Parents' Quality of Life | 6 months
  Parents' quality of life will be measured according to a subjective life appraisal definition with Diener's highly validated Satisfaction with Life Scale (SWLS) (5 items) which is the most validated life satisfaction scale in health and social sciences literature.
Parents' Quality of Life | 6 months
  Parents' quality of life will also be measured with an adapted version of the KIDSCREEN survey subscale for Feelings.
Parents' Quality of Life | 12 months
  Parents' quality of life will be measured according to a subjective life appraisal definition with Diener's highly validated Satisfaction with Life Scale (SWLS) (5 items) which is the most validated life satisfaction scale in health and social sciences literature.
Parents' Quality of Life | 24 months
  Parents' quality of life will be measured according to a subjective life appraisal definition with Diener's highly validated Satisfaction with Life Scale (SWLS) (5 items) which is the most validated life satisfaction scale in health and social sciences literature.
Parents' Quality of Life | 12 months
  Parents' quality of life will also be measured with an adapted version of the KIDSCREEN survey subscale for Feelings.
Parents' Quality of Life | 24 months
  Parents' quality of life will also be measured with an adapted version of the KIDSCREEN survey subscale for Feelings.
Parents' Perceived Emotional and Physical Health | Baseline
  Parents' perceived health, energy, and fatigue will be assessed with short forms of the Patient Reported Outcomes Measurement Information System (PROMIS).
Parents' Perceived Emotional and Physical Health | 6 months
  Parents' perceived health, energy, and fatigue will be assessed with short forms of the Patient Reported Outcomes Measurement Information System (PROMIS).
Parents' Perceived Emotional and Physical Health | 12 months
  Parents' perceived health, energy, and fatigue will be assessed with short forms of the Patient Reported Outcomes Measurement Information System (PROMIS).
Parents' Perceived Emotional and Physical Health | 24 months
  Parents' perceived health, energy, and fatigue will be assessed with short forms of the Patient Reported Outcomes Measurement Information System (PROMIS).
Effects of Child's Condition on Parents' Finances and Ability to Work | Baseline
  Financial Impact on Parents' will be measured using an Expense Diary survey created by the co-investigators.
Effects of Child's Condition on Parents' Finances and Ability to Work | 6 months
  Financial Impact on Parents' will be measured using an Expense Diary survey created by the co-investigators.
Effects of Child's Condition on Parents' Finances and Ability to Work | 12 months
  Financial Impact on Parents' will be measured using an Expense Diary survey created by the co-investigators.
Effects of Child's Condition on Parents' Finances and Ability to Work | 24 months
  Financial Impact on Parents' will be measured using an Expense Diary survey created by the co-investigators.

OTHER OUTCOMES:
Health systems outcomes | Baseline
  The investigators will link the patient-reported evaluation of the CCKO initiative with encoded health administrative data housed at ICES for consenting participants.
Health systems outcomes | 6 months
  The investigators will link the patient-reported evaluation of the CCKO initiative with encoded health administrative data housed at ICES for consenting participants.
Health systems outcomes | 12 months
  The investigators will link the patient-reported evaluation of the CCKO initiative with encoded health administrative data housed at ICES for consenting participants.
Health systems outcomes | 24 months
  The investigators will link the patient-reported evaluation of the CCKO initiative with encoded health administrative data housed at ICES for consenting participants.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Cohen, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (4):
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Cohen E, Quartarone S, Orkin J, Moretti ME, Emdin A, Guttmann A, Willan AR, Major N, Lim A, Diaz S, Osqui L, Soscia J, Fu L, Gandhi S, Heath A, Fayed N. Effectiveness of Structured Care Coordination for Children With Medical Complexity: The Complex Care for Kids Ontario (CCKO) Randomized Clinical Trial. JAMA Pediatr. 2023 May 1;177(5):461-471. doi: 10.1001/jamapediatrics.2023.0115. PMID 36939728
- [Derived] Orkin J, Chan CY, Fayed N, Lin JLL, Major N, Lim A, Peebles ER, Moretti ME, Soscia J, Sultan R, Willan AR, Offringa M, Guttmann A, Bartlett L, Kanani R, Culbert E, Hardy-Brown K, Gordon M, Perlmutar M, Cohen E. Complex care for kids Ontario: protocol for a mixed-methods randomised controlled trial of a population-level care coordination initiative for children with medical complexity. BMJ Open. 2019 Aug 1;9(8):e028121. doi: 10.1136/bmjopen-2018-028121. PMID 31375613